CLINICAL TRIAL: NCT03468075
Title: A Phase II Trial of Gemcitabine Plus High-Dose Ascorbate in Locally Advanced Unresectable or Metastatic Soft Tissue and Bone Sarcomas in Adults
Brief Title: Gemcitabine Plus Ascorbate for Sarcoma in Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopping rules met
Sponsor: Mohammed Milhem, MBBS (Other)
Collaborators: University of Iowa (Other); St. Baldrick's Foundation (Other)
Responsible Party: Principal Investigator, Varun Monga, MD, Assistant Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201802800 (Phase II)
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Sarcoma; Soft Tissue Sarcoma; Unresectable Soft Tissue Sarcoma; Metastatic Bone Tumor; Bone Sarcoma
Keywords: Sarcoma; Soft tissue; Ascorbate
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Ascorbic Acid; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + High-Dose Ascorbate (Experimental): Subjects will receive ascorbate, 75g, on Days 1, 2, 8, 9, 15 and 16 of a 28-day cycle. Gemcitabine will be administered on Days 1, 8 and 15, after the infusion of ascorbate. Concomitant treatment will continue for 6 cycles. Patients whose disease has not progressed while receiving gemcitabine and ascorbate and who are tolerating therapy may continue either single agent gemcitabine or concomitant treatment beyond 6 cycles at the discretion of the investigator.
  Interventions: Drug: Ascorbate; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbate — Following 15g test dose, 75g administered on Days 1, 2, 8, 9, 15 and 16 of a 28-day cycle
  Other Names: Ascorbic Acid; Vitamin C; Pharmacological ascorbate
Drug: Gemcitabine — Administered on Days 1, 8 and 15, after the infusion of ascorbate
  Other Names: Gemzar

SUMMARY:
This study will enroll patients who have a diagnosis of locally advanced, unresectable or metastatic soft tissue or bone sarcoma (except gastrointestinal stromal tumors and Kaposi's sarcoma) from any site.

DETAILED DESCRIPTION:
This study will enroll male and female patients 18 years old or older who have a diagnosis of locally advanced, unresectable or metastatic soft tissue or bone sarcoma (except GIST and Kaposi's) from any site. A minimum of 1 prior chemotherapy regimen, including adjuvant and neo-adjuvant therapy for the treatment of sarcoma, must have been given. Patients eligible for an anthracycline should have received a prior anthracycline containing regimen. Patients who decline or are not eligible for anthracycline treatment may be considered for this protocol as a first line treatment. Patients with a diagnosis of liposarcoma should also have received eribulin.

During screening, subjects will receive a test dose (15g) of ascorbate. If the test dose results in any toxicity >/= CTCAE grade 3 or a significant medical event in the opinion of the principal investigator, the patient will be considered a screen failure.

Subjects who pass screening will then receive ascorbate, 75g, on Days 1, 2, 8, 9, 15 and 16 of a 28-day cycle. Gemcitabine will be administered on Days 1, 8 and 15, after the infusion of ascorbate. Concomitant treatment will continue for at least 6 cycles. Patients whose disease has not progressed while receiving gemcitabine and ascorbate and who are tolerating therapy may continue either single agent gemcitabine or concomitant treatment beyond 6 cycles at the discretion of the investigator. Treatment will be terminated with progression of disease. Disease will be assessed by CT of the chest, abdomen and pelvis or MRI of the lesion every 2 cycles for progression.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old
2. ECOG Performance Status of ≤ 2
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed

   * Patients must meet the following laboratory criteria:
   * Hematology:
   * Neutrophil count of >1500/mm3
   * Platelet count of > 100,000/mm3L
   * Hemoglobin ≥ 9 g/dL (transfusion to meet eligibility allowed)
   * Biochemistry:
   * AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
   * Alkaline phosphatase < 5 x ULN
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
   * Total serum calcium >/= LLN or if calcium is below LLN then corrected calcium for serum albumin should be >/= LLN
   * Serum potassium ≥ LLN
   * Serum sodium ≥ LLN
   * Serum albumin ≥ LLN or 3g/dl
4. Tolerate a 15g ascorbate infusion (screening dose)
5. Baseline MUGA or ECHO done only in subjects with prior doxorubicin exposure. The test must demonstrate LVEF ≥ the lower limit of the institutional normal.
6. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
7. Any patient with the diagnosis of locally advanced, unresectable or metastatic soft tissue or bone sarcoma (except GIST and Kaposi's) from any site. A minimum of 1 prior chemotherapy regimen, including adjuvant and neo-adjuvant therapy for the treatment of sarcoma. Patients eligible for an anthracycline should have received a prior anthracycline containing regimen. Patients who decline or are not eligible for anthracycline treatment may be considered for this protocol as a first line treatment. Patients with a diagnosis of liposarcoma should also have received eribulin if they received anthracycline-based therapy prior to eribulin. Patients with a diagnosis of myxoid liposarcoma should have received trabectedin. Patients with angiosarcoma should have received either taxol or docetaxel. Patients must have measurable disease defined as at least 1 lesion ≥ 1cm in the greatest dimension.
8. Patients with metastatic bone sarcomas who have failed all available therapies that have demonstrated clinical benefit. Available therapies include but not limited to methotrexate, adriamycin and cisplatin for osteosarcoma and vincristine, adriamycin and Cytoxan, ifosfamide, etoposide (VAC/IE)for Ewing's sarcoma.
9. Previous exposure to Gemcitabine will only be allowed if there is no residual toxicity from previous treatments. Toxicity must be graded as 0 or 1 prior to study.
10. Patients must have had disease progression on or following their most recent treatment regimen or on presentation for the first time with locally advanced unresectable or metastatic disease.

Exclusion Criteria:

1. G6PD (glucose-6-phosphate dehydrogenase) deficiency
2. New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
3. History of myocardial infarction or unstable angina within 6 months prior to Day 1
4. History of stroke or transient ischemic attack within 6 months prior to Day 1
5. Known CNS disease, except for treated brain metastasis: Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
6. Actively receiving insulin or requiring fingerstick glucose monitoring at time of ascorbate infusion (unless an exception is granted by the IND sponsor, medical monitor, and the PI).
7. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
8. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
9. Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in subjects of child-bearing potential
10. Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide. High dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs.
11. Other concurrent severe and/or uncontrolled medical conditions
12. Patients who have received chemotherapy or any investigational drug < 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
14. Concomitant use of any anti-cancer therapy or radiation therapy. Palliative radiation therapy to non-target lesions is permitted.
15. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
16. Patients with a history of another primary malignancy within 2 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
17. Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required. High-dose ascorbate acid is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral drugs.
18. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
19. Patients with GIST tumors and Kaposi's Sarcoma are excluded.
20. Patients with history of more than one symptomatic oxalate stone in the last 6 months or visible stone in the kidney or ureter on screening CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2020-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varun Monga, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine + High-Dose Ascorbate
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + High-Dose Ascorbate
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 68 [52 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: From first day of treatment to documented disease progression as described by RECIST 1.1 criteria. Results are provided in nominal categories (CR, PR, SD, PD) as per RECIST.
Time Frame: Every 2 months for first 6 months, then every 3 months up to 2 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + High-Dose Ascorbate
Number analyzed (Participants) | 10
Participants
  PD | 8
  SD | 1
  PR | 1

2. Secondary Outcome: Progression Free Survival
Description: Time from start of therapy (day 1, cycle 1) to documented disease progression or death due to any cause. Progression will be defined using the RECIST 1.1 guidelines. Results are provided in nominal categories (CR, PR, SD, PD) as per RECIST.
Time Frame: Every 2 months for first 6 months, then every 3 months up to 2 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + High-Dose Ascorbate
Number analyzed (Participants) | 10
Participants
  2 months | 7
  3 months | 1
  6 months | 1
  9 months | 1

3. Secondary Outcome: Overall Survival
Description: Time from start of therapy (day 1, cycle 1) to death.
Time Frame: Every 2 months for first 6 months, then every 3 months up to 2 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine + High-Dose Ascorbate
Number analyzed (Participants) | 10
Participants
  Alive | 5
  Dead | 5

4. Secondary Outcome: Incidence of Adverse Events (AE) Per CTCAE 4.03
Description: Categorize and quantify adverse events from start of therapy (day 1, cycle 1) to end of study per (CTCAE) version 4.03.
Time Frame: Up to 30 days after completion of study treatment
Measure: Number; unit: adverse events
Arm/Group | Gemcitabine + High-Dose Ascorbate
Number analyzed (Participants) | 10
adverse events
  Blood and lymphatic system disorders | 4
  Gastrointestinal disorders | 7
  Infections and infestations | 1
  Investigations | 43
  Metabolism and nutrition disorders | 2
  Musculoskeletal and connective tissue disorders | 1
  Psychiatric disorders | 1
  Renal and urinary disorders | 1
  Respiratory, thoracic and mediastinal disorders | 11
  Skin and subcutaneous tissue disorders | 3
  Vascular disorders | 2
  General disorders and administration site conditions | 7

ADVERSE EVENTS:
Time Frame: AEs were collected up to 30 days after completion of study treatment, up to 7 months
Description: Information about all adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, were collected and recorded and followed as appropriate. Adverse events were followed for 30 days post last dose of drug.
Arm/Group | Gemcitabine + High-Dose Ascorbate
All-Cause Mortality (participants affected / at risk) | 6/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + High-Dose Ascorbate (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + High-Dose Ascorbate (N=10)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (3)
Pain (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 6 (9)
Platelet count decreased (Investigations) | 6 (26)
Weight loss (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Study terminated early. Ten patients were enrolled in the first stage, and per protocol the study was terminated following interim analysis when 1 or fewer participants had a tumor response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT03468075/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03468075/ICF_001.pdf